CLINICAL TRIAL: NCT02939950
Title: A Study to Evaluate the Safety and Effectiveness of a Silicone Hydrogel Soft Contact Lens When Worn on a 7-Day Extended Wear Basis
Brief Title: Silicone Hydrogel Soft Contact Lens 7-Day Extended Wear Basis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 818
Record Dates: First submitted 2015-06-01; First posted 2016-10-20 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch + Lomb Samfilcon A Soft Contact Lens (Experimental): Participants will wear Bausch + Lomb samfilcon A soft contact lens in each eye on a 7-day extended daily wear basis for a period of 12 months. The lenses will be worn overnight for up to 6 consecutive nights per week. The lenses will be removed, cleaned, and disinfected with Biotrue multi-purpose solution on the seventh night and re-inserted the following morning. The lenses will be replaced with new lenses on the first monday of each month.
  Interventions: Device: Bausch + Lomb Samfilcon A Soft Contact Lens
- Bausch + Lomb Pure Vision Soft Contact Lens (Active Comparator): Participants will wear Bausch + Lomb pure vision soft contact lens in each eye on a 7-day extended daily wear basis for a period of 12 months. The lenses will be worn overnight for up to 6 consecutive nights per week. The lenses will be removed, cleaned, and disinfected with Biotrue multi-purpose solution on the seventh night and re-inserted the following morning. The lenses will be replaced with new lenses on the first monday of each month.
  Interventions: Device: Bausch + Lomb Pure Vision Soft Contact Lens

INTERVENTIONS:
Device: Bausch + Lomb Samfilcon A Soft Contact Lens — soft contact lenses
  Arms: Bausch + Lomb Samfilcon A Soft Contact Lens
Device: Bausch + Lomb Pure Vision Soft Contact Lens — soft contact lenses
  Arms: Bausch + Lomb Pure Vision Soft Contact Lens

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Bausch + Lomb samfilcon A soft (hydrophilic) contact lens, a new silicone hydrogel contact lens, compared to the Bausch + Lomb PureVision® soft contact lens when worn for 7-day extended wear by adapted soft contact lens wearers.

DETAILED DESCRIPTION:
Approximately 816 participants (1,632 eyes) will be enrolled in this 12-month randomized, parallel, Investigator/Sponsor masked study at approximately 35 investigative sites in the US.

At the Screening/Dispensing Visit, approximately one-half of the participants will be randomized to receive Bausch + Lomb investigational samfilcon A soft contact lenses (Test) and approximately one-half of the subjects will be randomized to receive Bausch + Lomb PureVision soft contact lenses (Control). Both groups will wear the assigned lenses bilaterally on a 7-day extended wear basis throughout the 12 month study. The lenses are to be worn overnight for up to six consecutive nights per week. The lenses are to be removed, cleaned and disinfected on the seventh night and re-inserted the following morning. The lenses will be replaced with new lenses at the beginning of each month. Lenses will be provided at the Screening/Dispensing, 3-Month, 6-Month and 9-Month Follow-Up visits to maintain a monthly replacement schedule. Participants will also be required to complete a paper diary.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be correctable through spherocylindrical refraction to 42 letters (0.1 logMAR) or better (distance, high contrast) in each eye.
* Participants must be adapted lens wearers and wear a lens in each eye; each lens must be of the same manufacturer and brand.
* Participants must be myopic and require lens correction from -0.50 diopters (D) to 6.00 D in each eye.
* Participants must have clear central corneas and be free of any anterior segment disorders.
* Participants must agree to wear their lenses on an extended wear basis (6 nights/7 days) for the duration of the study.

Exclusion Criteria:

* Participants who have worn gas permeable (GP) contact lenses within the last 30 days or who have worn polymethylmethacrylate (PMMA) lenses within the last three months.
* Participants with an active ocular disease or who are using any ocular medication.
* Participants with any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study.
* Participants using any systemic medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Participants who are not correctable to 42 letters (0.1 logMAR) in each eye with soft spherical contact lenses.
* Participants who currently wear monovision, multifocal, or toric contact lenses.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 816 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Cicero Family Eye Care, Cicero, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1632 eyes from 816 study participants were enrolled, of which 1612 eyes from 806 study participants were randomized into 1:1 to wear either the Bausch + Lomb samfilcon A soft contact lens or Bausch + Lomb pure vision soft contact lens.
Units Other Than Participants: Eyes
Groups:
- Bausch + Lomb Samfilcon A Soft Contact Lens: Participants wore Bausch + Lomb samfilcon A soft contact lens in each eye on a 7-day extended daily wear basis for a period of 12 months. The lenses were worn overnight for up to 6 consecutive nights per week. The lenses were removed, cleaned, and disinfected with Biotrue multi-purpose solution on the seventh night and re-inserted the following morning. The lenses were replaced with new lenses on the first monday of each month.
- Bausch + Lomb Pure Vision Soft Contact Lens: Participants wore Bausch + Lomb pure vision soft contact lens in each eye on a 7-day extended daily wear basis for a period of 12 months. The lenses were worn overnight for up to 6 consecutive nights per week. The lenses were removed, cleaned, and disinfected with Biotrue multi-purpose solution on the seventh night and re-inserted the following morning. The lenses were replaced with new lenses on the first monday of each month.
Period: Overall Study
Arm/Group | Bausch + Lomb Samfilcon A Soft Contact Lens | Bausch + Lomb Pure Vision Soft Contact Lens
Started | 406; 812 Eyes | 410; 820 Eyes
Dispensed the Assigned Lenses | 405; 810 Eyes | 410; 820 Eyes
Eligible at Baseline | 403; 806 Eyes | 402; 804 Eyes
Completed | 340; 680 Eyes | 329; 658 Eyes
Not Completed | 66; 132 Eyes | 81; 162 Eyes
Not completed — Lost to Follow-up | 13 | 16
Not completed — Positive slit lamp findings | 0 | 1
Not completed — Chalazion upper lid | 0 | 1
Not completed — Lack of motivation | 0 | 2
Not completed — Unacceptable distance lens visual acuity | 1 | 1
Not completed — Military orders | 1 | 0
Not completed — Participant Relocated | 5 | 3
Not completed — Study related symptoms | 8 | 8
Not completed — Unacceptable lens movement | 2 | 0
Not completed — Protocol Violation | 6 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 6 | 7
Not completed — Withdrawal by Subject | 12 | 28
Not completed — Adverse Event | 7 | 3
Not completed — Randomized, not dispensed | 1 | 0
Not completed — Ineligible at Baseline | 2 | 8

BASELINE CHARACTERISTICS:
Population: Analysis set included all eligible dispensed participants under the treatment they actually received.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Bausch + Lomb Samfilcon A Soft Contact Lens | Bausch + Lomb Pure Vision Soft Contact Lens | Total
Number analyzed (Participants) | 403 | 402 | 805
Number analyzed (Eyes) | 806 | 804 | 1610
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (6.2) | 29.2 (6.1) | 29.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 265 | 528
  Male | 140 | 137 | 277

OUTCOME MEASURES:

1. Primary Outcome: High Contrast Visual Acuity
Description: For determination of high contrast visual acuity (VA), the participant was seated at the photoropter so that the distance from the participant's eyes to the logMAR chart was 6.5 feet (2.0 meters). The chart was at eye level for each participant. The logMAR charts had two alternative letter sequences from 28 letters (0.3 logMAR) to 62 letters (-0.3 logMAR). The visual acuity was measured through the phoropter using the distance refractive correction with the addition of +0.50 Diopter to compensate for the reduced test distance of 6.5 feet (2.0 meters). A scoring sheet for each eye was provided to keep track of the letters correctly identified by the participants. Scores were recorded as the numbers of letters correctly identified in the eye examination. VA was converted to the Log10 of the Minimum Angle of Resolution (logMAR) by using the score (number of letters).
Time Frame: Month 12
Population: Analysis set included all eligible dispensed participants under the treatment they actually received. Here, Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Bausch + Lomb Samfilcon A Soft Contact Lens | Bausch + Lomb Pure Vision Soft Contact Lens
Number analyzed (Participants) | 335 | 326
Number analyzed (eyes) | 669 | 652
logMAR | -0.065 (0.067) | -0.047 (0.071)

2. Primary Outcome: Number of Participants With Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events were defined as those events that resulted in, or had the potential to cause, either permanent impairment of an ocular function or damage to an ocular structure, and might necessitate medical or surgical intervention. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in reported AE section.
Time Frame: Baseline up to Month 12
Population: Safety analysis set included all dispensed participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Bausch + Lomb Samfilcon A Soft Contact Lens | Bausch + Lomb Pure Vision Soft Contact Lens
Number analyzed (Participants) | 405 | 410
Participants | 22 | 14

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: Safety analysis set included all dispensed participants. Participants were analyzed as treated. AEs related to eye were only recorded by investigators and no coding dictionary was used.
Arm/Group | Bausch + Lomb Samfilcon A Soft Contact Lens | Bausch + Lomb Pure Vision Soft Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/405 | 0/410
Serious Adverse Events (participants affected / at risk) | 0/405 | 0/410
Other Adverse Events (participants affected / at risk) | 22/405 | 14/410
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bausch + Lomb Samfilcon A Soft Contact Lens (N=405) | Bausch + Lomb Pure Vision Soft Contact Lens (N=410)
Peripheral Non-Progressive Non-Infectious Corneal Ulcer (Eye disorders) | 3 | 3
Symptomatic Corneal Infiltrative Event (Eye disorders) | 15 | 4
Corneal Staining greater than or equal to Grade 3 (Eye disorders) | 4 | 3
Ocular Event that necessitates temporary lens discontinuation for atleast two weeks (Eye disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.